CLINICAL TRIAL: NCT02617823
Title: Influence of Maternal Postioning on Spread of Local Anesthetic After Epidural Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Peter Bansch, Consultant Anesthetist, Region Skane
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SUSAN-KK
Record Dates: First submitted 2015-11-24; First posted 2015-12-01 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Effects of; Anesthesia, Spinal and Epidural, in Pregnancy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- semi-recumbent (No Intervention): rutine positioning at the hospital today
- lateral position (Experimental): experimental position to be evaluated against rutine
  Interventions: Procedure: lateral position

INTERVENTIONS:
Procedure: lateral position — patients placed on their left side after epidural catheter insertion
  Arms: lateral position

SUMMARY:
The purpose of this study is to determine if a lateral positioning of the pregnant woman after epidural analgesia increases the incidence of unilateral functioning epidurals.

DETAILED DESCRIPTION:
Pregnant women requesting epidural analgesia will be randomized to either left lateral or semi-recumbent position for 30 minutes after the first epidural bolus-injection.

After 30 minutes, the clinical effect of the analgesia will be evaluated by an anesthesiologist if available or by a midwife if the anesthesiologist is unavailable. The study-period is concluded thereafter and further positioning is optional.

Maternal and fetal wellbeing are continuously being monitored during the study period and complications/interventions registered. APGAR and CTG results during the intervention will be registered and evaluated at a later stage.

ELIGIBILITY:
Inclusion Criteria:

* all adult pregnant women recieiving epidural analgesia

Exclusion Criteria:

* participation refused
* inability to understand study purpose/instructions
* study postition could not be maintained for 30 min
* ineffective epidural

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 950 (Actual)
Dates: Start 2016-01; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
unilateral analgesic effect | evaluation of epidural effect after 30 min
  clinical judgement: mothers pain-sensation and cold sensation test

SECONDARY OUTCOMES:
maternal comfort and safety in regards to blood pressure and/or unexpected neurological effects from epidural analgesia | evaluation of epidural effect after 30 min
  clinical judgement: mothers subjective wellbeing, bloodpressure and incidence of vena cava compression, neurological deficits from epidural
fetal/neonatal safety measured with CTG and APGAR score | CTG from start of study until birth, APGAR 2, 5 and 10min after birth
  cardiotocographic changes and APGAR-score evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Samuelsson, MD, PhD, Study Chair — Region Skane, Head of the Department of Anesthesia and Intensive Care, University Hospital SUS
Locations (2):
- Sweden (2):
  - University Hospital SUS, Lund, Skåne County
  - University Hospital SUS, Malmo, Skåne County

IPD SHARING:
Plan to Share IPD: No